CLINICAL TRIAL: NCT05548023
Title: Time-trend Analysis of Clinical Characteristic and Outcomes in Patients With Unprotected Left Main Coronary Artery Disease Treated With PCI Over a 10-year Period
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023.464
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- unprotected left main coronary artery disease treated with PCI (Other)
  Interventions: Device: The AngioliteTM Durable Fluoroacrylate Polymer-based Sirolimus-Eluting Stent

INTERVENTIONS:
Device: The AngioliteTM Durable Fluoroacrylate Polymer-based Sirolimus-Eluting Stent — The Angiolite stent is a thin-strut cobalt-chromium sirolimus-eluting stent with an open-cell design and a high overexpansion capacity that might overcomes some of these challenges in LMCA PCI. The ANGIOLITE randomized trial confirmed the non-inferiority of the Angiolite stent against the conventional DES

SUMMARY:
Surgical coronary bypass surgery (CABG) has been demonstrated to confer significant survival benefit over medical therapies patients with LMCA in earlier clinical trials1,2,3 and therefore was the revascularization modality of choice for a long time. Recently, several randomized controlled trials and meta-analyses have shown percutaneous coronary intervention (PCI) to be non-inferior to CABG in the treatment of LMCA disease4,5,6,7,8. PCI is now considered to be an appropriate alternative to CABG for LMCA disease in patients with suitable anatomy9,10. Over recent decades, LMCA PCI has been performed in patients with increasing anatomical complexity and higher risk profiles (e.g. elderly, heart failure, renal failure etc). 11,12. In recent years, remarkable advancement in interventional techniques and technologies such as 2nd/3rd generation DES and potent antiplatelet therapy have contributed to the improvement of PCI success rates and reduction in complications and adverse events. Knowledge related to long term temporal variation of clinical and procedural characteristics and outcomes in patients with LMCA disease treated with PCI will therefore be important to inform and define future treatment strategies. This proposal aims to evaluate time-trends and regional differences in clinical characteristics and outcomes of patients with LMCA disease treated with PCI in the Asia-Pacific region

ELIGIBILITY:
Inclusion Criteria:

* Lp(a) ≥ 70 mg/dL at the screening visit
* Optimal LDL-cholesterol lowering treatment
* Optimal treatment of other CV risk factors
* Myocardial infarction: ≥ 3 months to ≤ 10 years prior to the screening visit, and/or
* Ischemic stroke: ≥ 3 months to ≤ 10 years prior to the screening visit, and/or
* Clinically significant symptomatic peripheral artery disease

Exclusion Criteria:

* Uncontrolled hypertension
* Heart failure New York Heart Association (NYHA) class IV
* History of malignancy of any organ system
* History of hemorrhagic stroke or other major bleeding
* Platelet count <140,000 per μL
* Active liver disease or hepatic dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2024-12-08 (Estimated); Study Completion 2025-02-07 (Estimated)

PRIMARY OUTCOMES:
Risk reduction of expanded MACE by TQJ230 | 51 months
  To demonstrate the superiority of TQJ230 compared to placebo in reducing the risk of expanded MACE (cardiovascular death, non-fatal MI, non-fatal stroke and urgent coronary re-vascularization requiring hospitalization) in 1) the overall study population with established CVD (Lp(a) ≥ 70 mg/dL) and/or 2) in a subpopulation with established CVD and Lp(a) ≥ 90 mg/dL.

SECONDARY OUTCOMES:
MACE reduction by TQJ230 | 51 months
  Demonstrate the superiority of TQJ230 compared to placebo in reducing the risk of the MACE composite of CV death, non-fatal MI and non-fatal stroke.
coronary heart disease (CHD) outcomes by TQJ230 | 51 months
  Demonstrate the superiority of TQJ230 compared to placebo in reducing the risk of the composite of coronary heart disease (CHD) outcomes: death due to CHD, non-fatal MI and urgent coronary re-vascularization requiring hospitalization. Evaluate the rate of all cause death.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Yan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong